CLINICAL TRIAL: NCT05159999
Title: The Home Blood Pressure (BP) Trial
Acronym: Home-BP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nisha Bansal, Associate Professor, Division of Nephrology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012367; R01DK123104 (NIH)
Record Dates: First submitted 2021-11-18; First posted 2021-12-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Blood pressure, dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Home Systolic Blood Pressure <140 mmHg (Experimental): Participants will take their home blood pressure two times per week (one in the morning and one in the evening) on non-dialysis days, ideally mid-week. Home blood pressures will be reviewed every two weeks and dry weight and medications adjusted accordingly to reach a home systolic blood pressure target of <140 mmHg.
  Interventions: Other: Dry weight target adjustment; Drug: Anti-hypertensive medications
- Pre-Dialysis Systolic Blood Pressure <140 mmHg (Active Comparator): Participants will have their blood pressure taken by an automated blood pressure device by dialysis unit staff using regular dialysis unit equipment according to usual clinical care. Pre-dialysis blood pressures will be reviewed every two weeks and dry weight and medications adjusted accordingly to reach a pre-dialysis systolic blood pressure target of <140 mmHg.
  Interventions: Other: Dry weight target adjustment; Drug: Anti-hypertensive medications
- Home Systolic Blood Pressure <130 mmHg (Other): This will be an optional, exploratory 2 month study at the end of the primary 10-month trial. Participants will take their home blood pressure two times per week (one in the morning and one in the evening) on non-dialysis days, ideally mid-week. Home blood pressures will be reviewed every two weeks and dry weight and medications adjusted accordingly to reach a home systolic blood pressure target of <130 mmHg.
  Interventions: Other: Dry weight target adjustment; Drug: Anti-hypertensive medications

INTERVENTIONS:
Other: Dry weight target adjustment — Target dry weight will be adjusted every 2 weeks to reach the home or pre-dialysis systolic blood pressure target.
Drug: Anti-hypertensive medications — Anti-hypertensive medications will be adjusted every 2 weeks to reach the home or pre-dialysis systolic blood pressure target. Adjustment of currently prescribed anti-hypertensive medications will be prioritized before starting new medications. Only standard anti-hypertensive medications will be used, such as RAAS inhibitors, beta-blockers, calcium channel blockers and diuretics.

SUMMARY:
The main study will be a two arm 10-month, cross-over randomized controlled trial of 200 participants treated with end-stage-kidney-disease treated with in-center hemodialysis in the Seattle and San Francisco area comparing a strategy of targeting home vs. pre-dialysis systolic blood pressure <140 mmHg to reduce rates of intradialytic hypotension. The target systolic blood pressure of <140 mmHg in both treatment groups will be achieved using an algorithm of dry weight adjustment and anti-hypertensive medication adjustment.

DETAILED DESCRIPTION:
The main study be a two arm 10-month, cross-over randomized controlled trial of 200 participants treated with in-center hemodialysis in the Seattle and San Francisco area comparing a strategy of targeting home vs. pre-dialysis systolic blood pressure <140 mmHg in reducing rates of intradialytic hypotension. The target systolic blood pressure of 100-140 mmHg will be achieved using an algorithm of volume management and anti-hypertensive medication adjustment every two weeks. Home blood pressure measures will be recorded throughout via a mobile health blood pressure monitor over the 10-month study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Undergoing in-center, thrice weekly hemodialysis for treatment of end stage renal disease (ESRD)
* Greater than 3 months since initiation of dialysis
* No anticipated change to peritoneal dialysis or kidney transplant within 10 months
* Life expectancy greater than 10 months
* Hypertension (defined as mean pre-dialysis SBP > 140 mmHg over prior 2 weeks or taking BP medications)
* Able to obtain/measure a brachial blood pressure at dialysis and at home (e.g., no left ventricular assist device, blood pressure not been taken routinely in lower extremity at dialysis unit)
* No condition that the primary nephrologist or PIs feel precludes participation

Exclusion Criteria:

* Incarcerated or institutionalized (prohibits home blood pressure measurement)
* Participating in another intervention study that may affect blood pressure
* Pregnant or anticipated pregnancy or breastfeeding (as this will require increase to more than three times a week dialysis and/or preclude use of some classes of blood pressure medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Intradialytic hypotension (IDH), defined as systolic blood pressure<90 mmHg during dialysis | 10 months
  Test the effect of treating home SBP <140mmHg vs a pre-dialysis SBP <140mmHg on rates of IDH

SECONDARY OUTCOMES:
Fatigue by SONG-HD Score | 10 months
  Test the effect of treating home SBP <140mmHg vs a pre-dialysis SBP <140mmHg on patient reported fatigue, as ascertained by the SONG-HD Fatigue Score (PMID: 33093215)
Cramping | 10 months
  Test the effect of treating home SBP <140mmHg vs a pre-dialysis SBP <140mmHg on frequency of cramping
Rates of hospitalizations for cardiovascular events and volume overload | 10 months
  Test the effect of treating home SBP <140mmHg vs a pre-dialysis SBP <140mmHg on rates of hospitalizations for cardiovascular events and volume overload
Correlation between pre-dialysis and home SBP | 10 months
  Evaluate the correlation between pre-dialysis and home SBP under different treatment strategies

OTHER OUTCOMES:
Separation of blood pressures | 2 months
  Determine whether the intervention is able to achieve a home systolic blood pressure <130mmHg in this optional study.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Bansal, MD, Principal Investigator — University of Washington; Chi-yuan Hsu, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided